CLINICAL TRIAL: NCT04932629
Title: A Proof of Concept Study to Evaluate the Clinical Safety and Efficacy of Ex-vivo Cultivated Allogenic Limbal Stem Cell Transplantation for Treatment of Superficial Corneal Pathologies".
Brief Title: To Evaluate the Clinical Safety and Efficacy of Limbal Stem Cell for Treatment of Superficial Corneal Pathologies".
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, Vivek Singh, Principal Investigator, L.V. Prasad Eye Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERF-SSC-SCP-01
Record Dates: First submitted 2021-02-17; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Corneal Scars and Opacities
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): The eligible patients will undergo corneal transplant surgery, when the central corneal epithelium will be removed using a surgical sponge. 0.1ml of stromal cells in a concentration of 0.5x106 cells/µl diluted in the thrombin component of fibrin glue (TISEEL, Baxter) will be applied to the debrided corneal stroma.
  Interventions: Biological: Ex-vivo cultivated Allogeneic limbal stromal stem cells

INTERVENTIONS:
Biological: Ex-vivo cultivated Allogeneic limbal stromal stem cells — n this prospective intervention study patients with unilateral superficial corneal scars will undergo a surgical procedure and in the second procedure, the eligible patients will undergo corneal transplant surgery, when the central corneal epithelium will be removed using a surgical sponge. 0.1ml of stromal cells in a concentration of 0.5x10*6 cells/µl diluted in the thrombin component of fibrin glue (TISEEL, Baxter) will be applied to the debrided corneal stroma. A soft bandage contact lens will be placed over the cornea at the end of the procedure. The patient will receive topical antibiotic and steroid eye drops in the post-operative period. Periodic comprehensive ophthalmic evaluation along with anterior segment optical coherence tomography (ASOCT) scanning and slit-lamp photography will be done at Day 1, Day 7, Day 30, Day 90, Day 180 and Day 360 and 720 Days post-surgery

SUMMARY:
This study proposes to investigate the transplantation of ex-vivo cultivated allogenic limbal stromal cells for the treatment of the corneal pathologies. The limbus is an ideal source as the stem cells are numerous and located very superficially in the tissue (17). Pre-clinical work suggests human corneal stromal stem cells can be isolated from the cadaveric tissues, cultivated in conditions suitable for cell based therapy and used to prevent fibrosis in a murine model of corneal stromal scarring. Further, these cells are able to successfully engraft, differentiate, and mediate wound healing in the corneal stroma such that the tissue remains healthy, free of fibrotic tissue, and optically transparent. The clinical implications of these findings are substantial in that it represents the potential to lessen the burden on donor tissue necessary for corneal allografts by using cultured cells to regenerate tissue. We foresee the ability of a clinician to and grow and expand the cells in number and after surgically removing the scar tissue from the wounded eye, apply the cultured limbal stem cells to regenerate healthy, transparent tissue.

DETAILED DESCRIPTION:
This would be a single-center prospective, open labeled, non-randomized interventional study. This study is an Investigator Initiated Study (IIS). The Ethics Committee of the LV Prasad Eye Institute, Hyderabad, would prospectively approve this study. This study would be conducted in strict adherence to the tenets of the Declaration of Helsinki, ICH GCP E6 (R2), Indian GCP Guidelines and New Drugs and Clinical Trial Rules 2019 and associated amendments and current National Ethical Guidelines for Biomedical and Health Research Involving Human Participants and Current National Stem Cell Research Guidelines and New Drugs and Clinical Trial Rules 2019.

Once the participants are found to be suitable for limbal transplant surgery, the patients will be administered written informed consent and audio /visual consent as per regulations. Detailed ophthalmic examination will be done to ensure that the patient is eligible for the trial.

All the screening procedures will be accomplished within 14± 7days. On Day 0 that is the date of surgery a Unique Participant Identification Number (UPIN) will be assigned to each patient and it would be in addition to hospital medical record number. The surgery will be done under local or general anesthesia (depending on age and patient preference).

In this prospective interventional study patients with unilateral superficial corneal scars will undergo a surgical procedure. Limbal ring from a cadaveric donor tissue, which is therapeutically accepted and serologically tested, is collected. This tissue will then be cultivated in the stem cell biology laboratory using standardized culture technique. Briefly the limbal tissue will be cut up into small pieces and digested overnight using an enzyme (Collagenase L). The cells obtained from the digest will be cultured on a petri-dish using 2% serum and growth factors. The cultured cells will be passaged three times to remove all epithelial cells from the culture.

In the second procedure, the eligible patients will undergo corneal transplant surgery, when the central corneal epithelium will be removed using a surgical sponge. 0.1ml of stromal cells in a concentration of 0.5x106 cells/µl diluted in the thrombin component of fibrin glue (TISEEL, Baxter) will be applied to the debrided corneal stroma. A soft bandage contact lens will be placed over the cornea at the end of the procedure. The patient will receive topical antibiotic and steroid eye drops in the post-operative period. Periodic comprehensive ophthalmic evaluation along with anterior segment optical coherence tomography (ASOCT) scanning and slit-lamp photography will be done at Day 1, Day 7, Day 30, Day 90, Day 180 and Day 360 and 720 Days post-surgery. The primary outcome measure of this study is to note any ocular or systemic adverse effects of this intervention at the various post-operative time points. The secondary outcome measures are visual improvement and change in the density and appearance of the corneal scarring and other pathologies after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants who are ≥18 and ≤ 60 years of age.
2. Patients having unilateral superficial corneal pathologies (defined as involving the anterior 200µM of the corneal stroma on ASOCT imaging)
3. Corneal burns, ulcers and scars
4. No prior history of corneal transplantation
5. No ongoing and other active ocular pathology
6. Candidate for stem cell transplant
7. No severe pathological and psychological conditions that might interfere with the patient's participation in the study
8. Able to provide written and audio-visual informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, for any reason without prejudice

Exclusion Criteria:

1. Bilateral corneal disease,
2. Corneal scars with limbal dysfunction (clinically defined as absent limbal palisades or conjunctivalization of the cornea)
3. Ocular surface disease including dry eye disease (defined as a Schirmer's test of less than 10mm at 5 minutes),
4. Unknown etiology, post-herpetic eye disease or eyes with active intra-ocular inflammation,
5. Children (<18 years of age),
6. Less than 3 months after documented clinical resolution of acute disease
7. Inability/refusal to give written informed consent
8. Undergo any of the anterior segment imaging tests.
9. Patient should have not participated in another clinical study within 30 days of their enrolment on this study.
10. History or evidence of cardiac disease: congestive heart failure; New York Heart Association (NYHA) class 2 or greater (see Appendix 6); active coronary artery disease; unstable angina, cardiac arrhythmias requiring anti-arrhythmic therapy, atrio-ventricular block of second or third degree, or uncontrolled hypertension, patients with recent (less than 6 months) myocardial infarction (MI) or coronary revascularization.
11. Pregnant and lactating patients, positive urine pregnancy test in women of childbearing potential
12. Reproductive age patients not practicing effective and adequate birth control measures
13. Previous participation in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of any ocular or systemic adverse effects | Day 90 post-surgery
  The primary outcome measure of this study is to note any ocular or systemic adverse effects

SECONDARY OUTCOMES:
Measurement of Visual improvement | Day 720 post surgery
  Visual improvement using ETDRS vision chart method where visual acuity is the measurement, Changes in ETDRS score is a scale and ETDRS letter score will be measure in log units
Change in Corneal light scattering | Day 720 post surgery
  Change in Corneal light scattering using Scheimpflug imaging where Corneal light scattering is the measurement, Corneal Densitometry measurements is a scale and expressed in standardized grayscale units (GSU).

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Vivek Singh, PhD, Principal Investigator — LV Prasad Eye Institute (Hyderabad Eye Research Foundation); Dr.Sayan Basu, MBBS.MS, Principal Investigator — LV Prasad Eye Institute (Hyderabad Eye Research Foundation)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basu S, Hertsenberg AJ, Funderburgh ML, Burrow MK, Mann MM, Du Y, Lathrop KL, Syed-Picard FN, Adams SM, Birk DE, Funderburgh JL. Human limbal biopsy-derived stromal stem cells prevent corneal scarring. Sci Transl Med. 2014 Dec 10;6(266):266ra172. doi: 10.1126/scitranslmed.3009644. PMID 25504883
- [Result] Basu S, Damala M, Singh V. Limbal Stromal Stem Cell Therapy for Acute and Chronic Superficial Corneal Pathologies: Early Clinical Outcomes of The Funderburgh Technique. Investigative Ophthalmology & Visual Science. 2017 Jun 23;58(8):3371-337
- [Result] Funderburgh, J., Basu, S., Damala, M., Tavakkoli, F., Sangwan, V., & Singh, V. (2018). Limbal stromal stem cell therapy for acute and chronic superficial corneal pathologies: one-year outcomes. Investigative Ophthalmology & Visual Science, 59(9), 3455-3455

DOCUMENTS (2):
  • Study Protocol (2019-03-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04932629/Prot_000.pdf
  • Informed Consent Form (2019-03-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04932629/ICF_001.pdf